CLINICAL TRIAL: NCT02475915
Title: A Randomized Study to Compare the Efficacy of Vorinostat/Hydroxychloroquine/Maraviroc (VHM) in Controlling HIV After Treatment Interruption in Subjects Who Initiated ART During Acute HIV Infection
Brief Title: Efficacy of VHM After Treatment Interruption in Subjects Initiating ART During Acute HIV Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SEARCH Research Foundation (Other)
Collaborators: The Thai Red Cross AIDS Research Centre (Unknown); Cooper Human Systems (Industry)
Responsible Party: Principal Investigator, Nitiya Chomchey, Prof.Praphan Phanuphak, MD, PhD, SEARCH Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEARCH 019
Record Dates: First submitted 2015-06-03; First posted 2015-06-19 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Acute HIV Infection
Keywords: Treatment interruption; Controlling HIV
MeSH Terms: interventions — Vorinostat; Hydroxychloroquine; Maraviroc; Tenofovir; Emtricitabine; efavirenz; Darunavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ART + VHM (Experimental): Group 1: Combination Antiretroviral Therapy prescribed at week 0 for a period of 10 weeks. Likely consisting of two NRTI such as tenofovir and emtricitabine and an NNRTI, such as efavirenz. For subjects on NNRTI therapy, a protease inhibitor, such as darunavir will be substituted for the NNRTI 2 weeks prior to treatment interruption.
  Plus: 3 X 14-day cycles of vorinostat administered at weeks 0, 4 and 8; hydroxychloroquine and maraviroc prescribed at week 0 for a period of 10 weeks.
  Interventions: Drug: Vorinostat; Drug: Hydroxychloroquine; Drug: Maraviroc; Drug: Tenofovir; Drug: Emtricitabine; Drug: Efavirenz; Drug: Darunavir
- ART alone (Active Comparator): Group 2: Combination Antiretroviral Therapy prescribed at week 0 for a period of 10 weeks. Likely consisting of two NRTI such as tenofovir and emtricitabine and either an NNRTI, such as efavirenz. For subjects on NNRTI therapy, a protease inhibitor, such as darunavir will be substituted for the NNRTI 2 weeks prior to treatment interruption.
  Interventions: Drug: Tenofovir; Drug: Emtricitabine; Drug: Efavirenz; Drug: Darunavir

INTERVENTIONS:
Drug: Vorinostat — Vorinostat (suberoylanilide hydroxamic acid) inhibits histone deacetylases class I and II. Vorinostat is supplied as 100mg capsules and will be administered at 400mg/ day in 2 week cycles beginning at week 0 for 10 weeks - 42 doses.
  Other Names: Zolinza
  Arms: ART + VHM
Drug: Hydroxychloroquine — Hydroxychloroquine is supplied as 200mg tablets and will be administered at week 0 for 10 weeks
  Other Names: Plaquenil
  Arms: ART + VHM
Drug: Maraviroc — Maraviroc will be administered at 150 to 600mg/ml twice daily depending on the subject's ART regimen at week 0 for 10 weeks
  Other Names: Selzentry
  Arms: ART + VHM
Drug: Tenofovir — NRTI. Tenofovir will be administered at 300mg 1 X day at week 0 for 10 weeks
  Other Names: Viread
Drug: Emtricitabine — NRTI. Emtricitabine will be administered at 200mg 1 X day at week 0 for 10 weeks
  Other Names: Emtriva
Drug: Efavirenz — NNRTI. Efavirenz will be administered at 600 mg 1 X day at week 0 for 10 weeks
  Other Names: Sustiva
Drug: Darunavir — Protease Inhibitor. Darunavir will be administered at a dose of 900mg 1 X day for subjects on NNRTI based ART beginning at week 8 until week 10
  Other Names: Prezista

SUMMARY:
This study is a two-arm prospective 1:1 randomised controlled trial comparing the proportion of patients between:

Group 1: vorinostat/hydroxychloroquine/maraviroc (VHM) co-administered with anti-retroviral therapy (ART) Group 2: ART only who are able to maintain HIV RNA < 50 copies/ml following treatment interruption. Subjects will be recruited from RV254/SEARCH 010, an acute HIV infection cohort conducted by the Thai Red Cross AIDS Research Centre in Bangkok, Thailand. The study will run for a minimum of 34 weeks from screening.

DETAILED DESCRIPTION:
Study site:

This will be a single-center proof-of-concept study in which recruitment and follow-up of volunteers will be done at the Thai Red Cross AIDS Research Centre (TRC-ARC).

Subject Population:

Subjects aged 18-60 years old, who initiated ART during acute HIV infection and have maintained viral suppression (HIV RNA < 50 copies/ml) for at least 28 weeks prior will be asked to enroll in the study. The subjects must have CD4 ≥ 450 cells/µl, and EKG and laboratory values within acceptable ranges.

Sample Size:

Fifteen subjects will be enrolled randomized 2:1 to VHM + ART (N=10) versus ART (N=5) only.

Study Design An exploratory, open label, randomized study of vorinostat/hydroxychloroquine/maraviroc (VHM) + ART versus ART only.

Study Drug Vorinostat will be administered at 400mg orally every 24h for 3 cycles, each of 14 days with an interim rest-period of 14 days between each cycle over a period of 10 weeks. Hydroxychloroquine (HCQ) will be administered at a dose of 200mg 2X/daily during the course of vorinostat administration for 10 weeks. Maraviroc will be administered at 600 mg 2X/daily on the same schedule as HCQ. This dose of maraviroc is based on its concomitant use with efavirenz. Dosing will be adjusted as appropriate should the subject be on an integrase inhibitor or a protease inhibitor instead of efavirenz due to intolerance to the drug or primary non-nucleoside reverse-transcriptase inhibitor (NNRTI) resistance. Any standard ART regimen may be used. However, it is expected that the majority of subjects will be on 2 nucleos(t)ide reverse-transcriptase inhibitors (NRTI) [emtricitabine (FTC) and tenofovir (TDF) and 1 NNRTI [efavirenz (EFV)]. ART will be administered at the following doses: FTC, 200mg 1X/day or 3TC, 300mg 1X/day; TDF, 300mg 1X/day and EFV, 600mg 1X/day.

In subjects on NNRTI-based therapy, the NNRTI will be interrupted at week 8 and the rest of the regimens will be interrupted at week 10. In order to prevent NNRTI resistance, protease inhibitor replacement therapy with darunavir (900 mg 1X/day with ritonavir 100 mg 1X/day) will be given between weeks 8 and 10 and maraviroc will be reduced from 1200mg/day to 300mg/day.

Study Duration on Protocol:

A minimum of 34 weeks from treatment initiation. Subjects must have been on ART for a minimum of 42 weeks prior to study entry. Note that some subjects may be enrolled from RV254/SEARCH010 who have already fulfilled the minimum 42-week ART requirement. The VHM treatment will occur over 10 weeks and the follow-up period will be 24 weeks.

Study Design and Methodology:

The study design is a two-arm, open label randomized study. Subjects will be recruited from RV254/SEARCH 010. RV254/SEARCH 010 is an acute HIV infection cohort conducted by the Thai Red Cross AIDS Research Centre in Bangkok, Thailand. Subjects will be followed twice daily for the first 24h following the first treatment administration and then at weeks 1, 2, 4, 5, 6, 8 and 10 and weekly thereafter to week 22, and every 2 weeks thereafter until week 34. Phlebotomy will be performed for clinical hematology, CD4, HIV RNA, ALT, creatinine and lipids and those in the VHM arm will also receive an EKG and eye examination at screening and/or enrollment. Subjects will be monitored weekly following treatment interruption for the following 12 weeks for viral load and every two weeks to week 34 to ensure that there is no viral rebound, defined as 2 consecutive viral load measurements of >1000 copies/ml. ART will be re-initiated and CD4 counts measured in the event of viral rebound.

A smaller proviral reservoir and less diverse viral population occur in early HIV infection relative to chronic infection. Preliminary data from the RV254/SEARCH 010 study indicate that T cell immunity is better preserved in subjects treated with ART during early HIV infection relative to chronic HIV infection.

The investigators hypothesize that subjects treated with ART during early HIV infection and further treated with multiple cycles of the histone deacetylase inhibitor (HDACi), vorinostat, in combination with hydroxychloroquine and maraviroc will lead to activation of the latent reservoir and reduce virus infection of new targets. Furthermore, as subjects were treated with ART early in HIV infection, the T cell response will be capable of eliminating virus activated by the HDACi and result in a reduction of the viral reservoir.

Primary Objective:

To compare the proportion of patients between VHM co-administered withART versus ART only arms who are able to maintain HIV RNA < 50 copies/ml following treatment interruption.

Secondary Objectives:

1. Time to HIV RNA rebound after treatment interruption between VHM +ART versus ART only arms
2. To compare the cell-associated HIV RNA (multi-spliced and unspliced) in total CD4+ T cells between the VHM +ART versus ART only arms
3. To compare markers of HIV persistence (total and integrated HIV DNA and 2-LTR circles) between the VHM + ART versus ART only arms
4. To compare histone acetylation (H3) between the VHM +ART versus ART only arms
5. To compare adverse events both related and unrelated to the combination of vorinostat, hydroxychloroquine and maraviroc between arms
6. To compare the occurrence and severity of acute retroviral syndrome between arms following treatment interruption

Hypotheses: Compared to the ART only arm, the VHM +ART arm will have:

1. A higher proportion of patients with HIV RNA < 50 copies/ml following treatment interruption at the end of the study
2. Longer time to HIV RNA rebound following treatment interruption
3. Higher cell-associated RNA in total CD4+ T cells at the end of the VHM treatment period
4. Lower reservoir size and 2 LTR circles at the end of the VHM treatment period and the end of the study
5. Higher histone acetylation at the end of the VHM treatment
6. Higher adverse events related to VHM
7. Similar rates of acute retroviral syndrome after treatment interruption in subjects experiencing viral rebound

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected adults 18-60 years
* Initiated ART during acute HIV infection period, defined serologically as up to a positive but incomplete profile by Western blot and has been on ART for at least 42 weeks
* HIV RNA <50 copies/ml within the past 7 months (28 weeks)
* CD4 cell count ≥ 450 cells/μl on at least 2 occasions during the past 6 months
* Informed consent

Exclusion Criteria:

* Any significant medical illness in the past 12 weeks
* Any evidence of AIDS-defining opportunistic infection
* Current or gastrointestinal disease that may impact absorption of the study drug
* ALT or AST >3X upper limit of normal
* Hemoglobin, white blood cell counts or platelets ≥ grade 2 by US NIH DAIDS grading system
* History of diabetes or fasting glucose >126mg/dl
* Documented hepatitis B infection as indicated by the presence of HBsAG
* History of clinically significant cardiac disease or clinically significant EKG abnormalities
* History of retinal disease
* History of malignancy
* Females who are pregnant or with a positive urine pregnancy test during screening or women of child bearing potential who are unwilling to use an acceptable method of contraception to avoid pregnancy for 4 weeks before, during the study and 4 weeks after the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with HIV RNA < 50 copies/ml following ART interruption | 24 weeks

SECONDARY OUTCOMES:
Time to HIV RNA rebound after treatment interruption between VHM +ART versus ART only arms defined as > 1000 HIV-1 RNA copies/ml on two consecutive plasma samples | 24 weeks
To compare the cell-associated spliced HIV RNA in total CD4+ T cells between the VHM+ ART and ART only arms. Measured as copies multi-spliced RNA/1000000 cells | 34 weeks
  HIV expression
To compare the cell-associated unspliced HIV RNA in total CD4+ T cells between the VHM+ ART and ART only arms. Measured as copies unspliced RNA/1000000 18S | 34 weeks
  HIV expression
To compare markers of HIV persistence measured as total, integrated and 2-LTR circles HIV DNA. Measured as DNA copies/1000000 cells | 34 weeks
  HIV persistence
To compare histone acetylation between the VHM + ART and ART only groups Expressed as mean fluorescence intensity | 10 weeks
  Serious Adverse Events
To compare adverse events both related and unrelated to the combination of hydroxychloroquine and maraviroc between arms graded according to NCI Common Terminology for Adverse Events | 34 weeks
  Serious Adverse Events
The occurrence and severity of acute retroviral syndrome between arms following treatment interruption using a combination of at least 3 clinical symptoms such as fever, lymphadenopathy and pharyngitis | 34 weeks
  Acute Retroviral Syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Somchai Sriplienchan, MD, MPH, Principal Investigator — SEARCH Research Foundation
Locations (1):
- SEARCH, the Thai Red Cross AIDS Research Centre, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schuetz A, Deleage C, Sereti I, Rerknimitr R, Phanuphak N, Phuang-Ngern Y, Estes JD, Sandler NG, Sukhumvittaya S, Marovich M, Jongrakthaitae S, Akapirat S, Fletscher JL, Kroon E, Dewar R, Trichavaroj R, Chomchey N, Douek DC, O Connell RJ, Ngauy V, Robb ML, Phanuphak P, Michael NL, Excler JL, Kim JH, de Souza MS, Ananworanich J; RV254/SEARCH 010 and RV304/SEARCH 013 Study Groups. Initiation of ART during early acute HIV infection preserves mucosal Th17 function and reverses HIV-related immune activation. PLoS Pathog. 2014 Dec 11;10(12):e1004543. doi: 10.1371/journal.ppat.1004543. eCollection 2014 Dec. PMID 25503054
- [Background] Ananworanich J, Schuetz A, Vandergeeten C, Sereti I, de Souza M, Rerknimitr R, Dewar R, Marovich M, van Griensven F, Sekaly R, Pinyakorn S, Phanuphak N, Trichavaroj R, Rutvisuttinunt W, Chomchey N, Paris R, Peel S, Valcour V, Maldarelli F, Chomont N, Michael N, Phanuphak P, Kim JH; RV254/SEARCH 010 Study Group. Impact of multi-targeted antiretroviral treatment on gut T cell depletion and HIV reservoir seeding during acute HIV infection. PLoS One. 2012;7(3):e33948. doi: 10.1371/journal.pone.0033948. Epub 2012 Mar 30. PMID 22479485
- [Background] Saez-Cirion A, Bacchus C, Hocqueloux L, Avettand-Fenoel V, Girault I, Lecuroux C, Potard V, Versmisse P, Melard A, Prazuck T, Descours B, Guergnon J, Viard JP, Boufassa F, Lambotte O, Goujard C, Meyer L, Costagliola D, Venet A, Pancino G, Autran B, Rouzioux C; ANRS VISCONTI Study Group. Post-treatment HIV-1 controllers with a long-term virological remission after the interruption of early initiated antiretroviral therapy ANRS VISCONTI Study. PLoS Pathog. 2013 Mar;9(3):e1003211. doi: 10.1371/journal.ppat.1003211. Epub 2013 Mar 14. PMID 23516360
- [Background] Elliott JH, Wightman F, Solomon A, Ghneim K, Ahlers J, Cameron MJ, Smith MZ, Spelman T, McMahon J, Velayudham P, Brown G, Roney J, Watson J, Prince MH, Hoy JF, Chomont N, Fromentin R, Procopio FA, Zeidan J, Palmer S, Odevall L, Johnstone RW, Martin BP, Sinclair E, Deeks SG, Hazuda DJ, Cameron PU, Sekaly RP, Lewin SR. Activation of HIV transcription with short-course vorinostat in HIV-infected patients on suppressive antiretroviral therapy. PLoS Pathog. 2014 Nov 13;10(10):e1004473. doi: 10.1371/journal.ppat.1004473. eCollection 2014 Oct. PMID 25393648
- [Background] Archin NM, Liberty AL, Kashuba AD, Choudhary SK, Kuruc JD, Crooks AM, Parker DC, Anderson EM, Kearney MF, Strain MC, Richman DD, Hudgens MG, Bosch RJ, Coffin JM, Eron JJ, Hazuda DJ, Margolis DM. Administration of vorinostat disrupts HIV-1 latency in patients on antiretroviral therapy. Nature. 2012 Jul 25;487(7408):482-5. doi: 10.1038/nature11286. PMID 22837004
- [Background] Bratland A, Dueland S, Hollywood D, Flatmark K, Ree AH. Gastrointestinal toxicity of vorinostat: reanalysis of phase 1 study results with emphasis on dose-volume effects of pelvic radiotherapy. Radiat Oncol. 2011 Apr 8;6:33. doi: 10.1186/1748-717X-6-33. PMID 21473790
- [Background] Chomont N, El-Far M, Ancuta P, Trautmann L, Procopio FA, Yassine-Diab B, Boucher G, Boulassel MR, Ghattas G, Brenchley JM, Schacker TW, Hill BJ, Douek DC, Routy JP, Haddad EK, Sekaly RP. HIV reservoir size and persistence are driven by T cell survival and homeostatic proliferation. Nat Med. 2009 Aug;15(8):893-900. doi: 10.1038/nm.1972. Epub 2009 Jun 21. PMID 19543283
- [Background] Abel S, Back DJ, Vourvahis M. Maraviroc: pharmacokinetics and drug interactions. Antivir Ther. 2009;14(5):607-18. PMID 19704163
- [Background] Ananworanich J, Hirschel B. Intermittent therapy for the treatment of chronic HIV infection. AIDS. 2007 Jan 11;21(2):123-34. doi: 10.1097/01.aids.0000256414.91105.8e. No abstract available. PMID 17197802
- [Background] Paton NI, Goodall RL, Dunn DT, Franzen S, Collaco-Moraes Y, Gazzard BG, Williams IG, Fisher MJ, Winston A, Fox J, Orkin C, Herieka EA, Ainsworth JG, Post FA, Wansbrough-Jones M, Kelleher P; Hydroxychloroquine Trial Team. Effects of hydroxychloroquine on immune activation and disease progression among HIV-infected patients not receiving antiretroviral therapy: a randomized controlled trial. JAMA. 2012 Jul 25;308(4):353-61. doi: 10.1001/jama.2012.6936. PMID 22820788
- [Background] Piconi S, Parisotto S, Rizzardini G, Passerini S, Terzi R, Argenteri B, Meraviglia P, Capetti A, Biasin M, Trabattoni D, Clerici M. Hydroxychloroquine drastically reduces immune activation in HIV-infected, antiretroviral therapy-treated immunologic nonresponders. Blood. 2011 Sep 22;118(12):3263-72. doi: 10.1182/blood-2011-01-329060. Epub 2011 May 16. PMID 21576701
- [Background] Prince HM, Bishton MJ, Harrison SJ. Clinical studies of histone deacetylase inhibitors. Clin Cancer Res. 2009 Jun 15;15(12):3958-69. doi: 10.1158/1078-0432.CCR-08-2785. Epub 2009 Jun 9. PMID 19509172
- [Background] Beliakova-Bethell N, Zhang JX, Singhania A, Lee V, Terry VH, Richman DD, Spina CA, Woelk CH. Suberoylanilide hydroxamic acid induces limited changes in the transcriptome of primary CD4(+) T cells. AIDS. 2013 Jan 2;27(1):29-37. doi: 10.1097/QAD.0b013e32835b3e26. PMID 23221426
- [Background] Lewin SR. A cure for HIV: where we've been, and where we're headed. Lancet. 2013 Jun 15;381(9883):2057-8. doi: 10.1016/S0140-6736(13)61180-0. No abstract available. PMID 23769215
- [Background] Katlama C, Deeks SG, Autran B, Martinez-Picado J, van Lunzen J, Rouzioux C, Miller M, Vella S, Schmitz JE, Ahlers J, Richman DD, Sekaly RP. Barriers to a cure for HIV: new ways to target and eradicate HIV-1 reservoirs. Lancet. 2013 Jun 15;381(9883):2109-17. doi: 10.1016/S0140-6736(13)60104-X. Epub 2013 Mar 29. PMID 23541541